CLINICAL TRIAL: NCT05591768
Title: The Clinical Efficacy of Monopolar Versus Bipolar Radiofrequency Ablation of the Genicular Nerves in the Treatment of Knee Osteoarthritis Pain.
Brief Title: Monopolar Versus Biopolar Radiofrequency in OA Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Abo Elkasem, principal investigatr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Radiofrequency in OA knee pain
Record Dates: First submitted 2022-08-18; First posted 2022-10-24 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBA group monopolar radiofrequency group. (Experimental): Inferomedial, superomedial, and superolateral GN branches of the patients were identified with ultrasonography, and a 22 Gauge, 10 cm radiofrequency (RF) cannula with a 10 mm active tip was advanced to the targeted nerves under fluoroscopy guidance. The location of the RF cannula was visualized by anteriorposterior and lateral images. Sensory stimulation was applied at 50 Hz to determine the nerve position. Since the sensory stimulation threshold must be < 0.6 V, nerve position was tested with the absence of fasciculation in the relevant area of the lower extremity upon 2.0 V stimulation at 2 Hz.
  Interventions: Procedure: Monopolar radiofrequency
- BFA group bipolar radiofrequency group (Experimental): similar technique will be used to insert the canula, except that, instead of one cannula two cannulae (approximately 10 mm apart) apart) will be inserted and no manipulation of cannulae was done to stimulate the target nerve as done in MRFA Target areas were similar to monopolar technique Each nerve will be ablated for 90 s in both the groups. All procedures were done by one pain physician who had more then 10 years' experience of radiofrequency procedures
  Interventions: Procedure: Bipolar radiofrequency

INTERVENTIONS:
Procedure: Monopolar radiofrequency — In monopolar group : . Inferomedial, superomedial, and superolateral GN branches of the patients were identified with ultrasonography, and a 22 Gauge, 10 cm radiofrequency (RF) cannula with a 10 mm active tip was advanced to the targeted nerves under fluoroscopy guidance. The location of the RF cannula was visualized by anteriorposterior and lateral images. Sensory stimulation was applied at 50 Hz to determine the nerve position. Since the sensory stimulation threshold must be < 0.6 V, nerve position was tested with the absence of fasciculation in the relevant area of the lower extremity upon 2.0 V stimulation at 2 Hz.
  Arms: MBA group monopolar radiofrequency group.
Procedure: Bipolar radiofrequency — a similar technique will be used to insert the canula, except that, instead of one cannula two cannulae (approximately 10 mm apart) apart) will be inserted and no manipulation of cannulae was done to stimulate the target nerve as done in MRFA Target areas were similar to monopolar technique Each nerve will be ablated for 90 s in both the groups. All procedures were done by one pain physician who had more then 10 years' experience of radiofrequency procedures.
  Arms: BFA group bipolar radiofrequency group

SUMMARY:
This is a prospective randomized controlled trial study will aim to evaluate the the efficacy and procedural pain of BRFA and to compare it with conventional technique (MRFA). And to compare the complications and time taken to complete the procedures.

DETAILED DESCRIPTION:
Chronic knee pain due to osteoarthritis (OA) is a debilitating disease. Many therapeutic options have been used to manage this pain . Although there are many pharmacological and surgical treatment options for knee osteoarthritis, these entail a number of concerns. Non-steroidal anti-inflammatory drugs can be used for the initial management of osteoarthritis . Intra-articular corticosteroid injection is another option suggested in the guidelines for the treatment of knee osteoarthritis . Surgical procedures are generally performed in cases unresponsive to the conservative treatment options. Joint replacement is the most commonly performed surgical procedure .Genicular nerve ablation with radiofrequency (RF) has recently become a promising treatment option in the management of osteoarthritis related knee pain. In conventional monopolar radiofrequency ablation (MRFA) technique, the localisation of genicular nerves is done through sensory stimulation at the junction of epicondyle with the shaft of femur bone near periosteum. Added to this, the procedure can be distressing when during localisation of genicular nerves the RF cannula comes in contact with pain-sensitive structures such as the periosteum and ligament insertion sites . Bipolar radiofrequency ablation Two radiofrequency cannula are advanced towards the nerve. The novel idea to use bipolar RFA in this study was to produce a larger lesion, thus may minimize the chance to miss the lesion of genicular nerves. Also Placing two electrodes avoids manipulation required to localise the genicular nerves with inadvertent stimulation of pain-sensitive periosteum . So investigaters need to see experimentally if bipolar radiofrequency ablation (BRFA) near the target nerve area without manipulation for localisation of genicular nerves has the ability to reduce the procedural pain than Monopolar radiofrequency.

ELIGIBILITY:
Inclusion Criteria:

* (1) outpatient clinic with osteoarthritis-character chronic knee pain, OA grades II-IV (Kellgren and Lawrence scale).

  (2) Patients not responding to other treatments as physiotherapy, oral analgesics, and intraarticular injection with hyaluronic acids or steroids.

  (3) Patients refused surgery. (4) Patients after failed conservative treatment for 3 months and reported more than 50% pain relief after diagnostic genicular nerve block with 2% of 2 mL lidocaine on superior lateral, superior medial and inferior medial genicular nerves.

Exclusion Criteria:

1. Patients with acute knee pain, previous knee surgery, other connective tissue disorders affecting the knee.
2. serious neurologic or psychiatric disorders, those had previously received radiofrequency ablation therapy for similar symptoms.
3. contraindications for genicular nerve block or genicular nerve RF (active infection, bleeding disorders, current use of anticoagulants or antiplatelets, allergy against the drugs used during the protocol, pregnancy, cardiac pacemaker.

   -

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy and procedural pain | Baseline
  Is to evaluate the efficacy and procedural pain of BRFA and to compare it with conventional technique (MRFA) by questionnaire participants

SECONDARY OUTCOMES:
Time | 2 years
  Is to compare time taken to complete the procedures

CONTACTS AND LOCATIONS:
Overall Officials: Hany Ahmed ibrahim, Professor, Study Chair — Assiut University
Locations (1):
- Assuit University hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi WJ, Hwang SJ, Song JG, Leem JG, Kang YU, Park PH, Shin JW. Radiofrequency treatment relieves chronic knee osteoarthritis pain: a double-blind randomized controlled trial. Pain. 2011 Mar;152(3):481-487. doi: 10.1016/j.pain.2010.09.029. Epub 2010 Nov 4. PMID 21055873
- [Background] Protzman NM, Gyi J, Malhotra AD, Kooch JE. Examining the feasibility of radiofrequency treatment for chronic knee pain after total knee arthroplasty. PM R. 2014 Apr;6(4):373-6. doi: 10.1016/j.pmrj.2013.10.003. Epub 2013 Dec 27. PMID 24373908